CLINICAL TRIAL: NCT00373269
Title: Procoagulant Effects of Hyperglycemia After Acute Stroke: A Pilot Study
Status: Completed | Type: Observational
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Other Study IDs: 3866 4187
Record Dates: First submitted 2006-09-05; First posted 2006-09-08 (Estimated); Results first posted 2017-01-04 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-01

CONDITIONS: Ischemic Stroke; Hyperglycemia
Keywords: Acute ischemic stroke; Stroke; Hyperglycemia; Procoagulation; Diabetes; Blood coagulation
MeSH Terms: conditions — Ischemic Stroke; Hyperglycemia; Stroke; Diabetes Mellitus; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diabetic subject: Subjects with acute stroke, hyperglycemia and history of diabetes.
- Normoglycemic Control: Subjects with acute stroke and normal blood glucose.

SUMMARY:
Between twenty and fifty percent of people who have acute stroke have hyperglycemia (high blood sugar) with it. The purpose of this study is to examine the relationships between diabetes mellitus, hyperglycemia,whole blood tissue factor procoagulant activity (TF-PCA) and plasma factorVIIa (FVIIa) in ten patients with type 2 diabetes mellitus and 11 non-diabetic patients at baseline and 6, 12, 24, and 48 hours (h) after presentation for acute stroke.

DETAILED DESCRIPTION:
The purpose of this study is to examine the relationships between diabetes mellitus, hyperglycemia,whole blood tissue factor procoagulant activity (TF-PCA) and plasma factorVIIa (FVIIa) in ten patients with type 2 diabetes mellitus and 11 non-diabetic patients at baseline and 6, 12, 24, and 48 hours (h) after presentation for acute stroke.

Patients presenting to the Emergency Department with ongoing stroke symptoms and neurologic deficit less than 24 hours (h) duration were screened for inclusion into the study. Stroke patients were grouped in terms of diabetes status as determined by past medical history. Stroke diagnosis was confirmed with brain magnetic resonance imaging (MRI). Clinical care, including the acute management ofstroke and hyperglycemia, was done at the discretion of the Neurology service not involved in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 years presenting to the Emergency Department with symptoms of acute ischemic stroke will be included for study.
* Acute stroke patients with normal blood glucose levels and patients with fingerstick blood glucose level of greater than or equal to 150 mg/dl will be eligible for study.
* Acute Stroke will be defined as an acute disturbance of cerebral function of presumed vascular origin causing a neurological deficit of less than 24 hours duration.
* Patients must have an NIH Stroke Scale Score of 4 to 23. Patients awakening with symptoms of stroke will be considered to have had their stroke at the time when last awake without symptoms.

Exclusion Criteria:

* Patients presenting after 24 hours of symptom onset. When the actual time of onset is unknown, the time when last observed to be symptom-free will be used.
* Patients with NIH scale of less than 4 or greater than 23.
* Complete or substantial resolution of symptoms before randomization.
* Patients with a previously disabling stroke (modified Rankin score > 3)
* Patients with other systemic disease such as infection (eg pneumonia, etc)
* Patients with hemorrhage visualized on CT.
* Patients who are unwilling or unable to give informed consent, or for whom a legally authorized representative is not able to consent.
* Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the Emergency Department with acute ischemic stroke within 12 hours of onset of symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2001-10; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina T Gentile, MD, Principal Investigator — Temple University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Normoglycemic Control: Subjects with acute ischemic stroke and normal blood glucose.
- Hyperglycemic Subjects: Subjects with acute ischemic stroke and hyperglycemia.
Period: Overall Study
Arm/Group | Normoglycemic Control | Hyperglycemic Subjects
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Normoglycemic: Subjects with acute ischemic stroke and normal blood glucose.
- Hyperglycemic: Subjects with acute ischemic stroke and hyperglycemia.
- Total: Total of all reporting groups
Arm/Group | Normoglycemic | Hyperglycemic | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 13
  >=65 years | 5 | 3 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (17.7) | 63.5 (9.2) | 64.2 (18.4)
Gender [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 6 | 3 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: FVIIa
Description: FVIIa levels were compared between the normoglycemic and hyperglycemic subjects.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mU/ml
Arm/Group | Normoglycemic Control | Hyperglycemic Subjects
Number analyzed (Participants) | 11 | 10
mU/ml | 69.7 (33.3) | 124.4 (35.2)

2. Secondary Outcome: TF-PCA
Description: TF-PCA levels compared between normoglycemic and hyperglycemic subjects.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: U/ml
Arm/Group | Normoglycemic Control | Hyperglycemic Subjects
Number analyzed (Participants) | 11 | 10
U/ml | 183.5 (63.1) | 118.1 (56.9)

ADVERSE EVENTS:
Description: Serious and Other (Not Including Serious) Adverse Events were not collected/assessed.
Arm/Group | Diabetic Subject | Normoglycemic Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes